CLINICAL TRIAL: NCT05272007
Title: Endoscopic Ultrasonography (EUS) Guided Gallbladder Drainage With Two Months Stent Removal for Acute Cholecystitis: a Prospective Study
Acronym: AC LAMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas Mater Domini (Other)
Responsible Party: Sponsor
Other Study IDs: 06-2022
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute cholecystitis
  Interventions: Procedure: EUS-biliary drainage

INTERVENTIONS:
Procedure: EUS-biliary drainage — EUS-GBD with LAMS

SUMMARY:
Acute cholecystitis (AC) is defined as an acute inflammatory disease of the gallbladder consequently to the presence of sludge or stones. AC accounts for 3-10% of all cases of abdominal pain. Cholecystolithiasis accounts for 90-95% of all causes of acute cholecystitis, while acalculous cholecystitis accounts for the remaining 5-10% of the cases. Laparoscopic cholecystectomy is actually the gold standard treatment for acute cholecystitis (AC) although it is always not suitable for patients who are poor candidates for surgery [ ]. In 2001 Giovannini et al. described the first EUS-guided biliary drainage (EUS-BD) through a transduodenal access with a needle knife. Subsequently, EUS-BD has considerably evolved thanks to the development of dedicated devices such as lumen apposing metal stents (LAMS), specifically designed for endoscopic ultrasound procedures. LAMS are made up of braided nitinol, that is fully covered with silicone to prevent tissue ingrowth, with wide flanges on both ends to provide anchorage.

Recently, LAMS have been incorporated into a delivery system with an electrocautery mounted on the tip which allows the device to be used directly to penetrate the target structure without the need to utilize a 19G needle, a guidewire, and a cystotome for prior dilation. Different are actually the indication of the LAMS for different disease and its use has been described for drainage of peri-pancreatic fluid collections, common bile duct (CBD), gallbladder, and for creation of gastro-jejuno anastomosis.

Recently, endoscopic gallbladder (GB) drainage was found to be a potentially revolutionary alternative for cholecystectomy for the control of symptoms, definitive treatment, or bridging therapy until surgery is possible.

Before the advent of LAMS, the standard of care of acute cholecystitis (AC) was the percutaneous drainage (PTC) and after the advent of these new stents, different series showed the higher technical and clinical success of the EUS-gallbladder drainage (EUS-GB) for acute cholecystitis, with a lower recurrence rate, than PTC. The superiority of this technique was assessed in terms of technical and clinical success, AEs and AC recurrence if compared to the endoscopic drainage. This could be explained with the use of larger caliber stents, allowing an effective drainage, with low risk of stent occlusion. Finally, a recent study with a long-term follow-up showed as the outcomes of EUS-GBD for AC were comparable with LC with acceptable rates of recurrent acute cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients arrived to the ER for AC with clinical and radiological evidence of AC (such as abdominal ultrasound, computed tomography or magnetic resonance)
* EUS gallbladder accessibility from the duodenum or from the stomach for the drainage
* Agree to receive follow up phone calls
* Able to provide written informed consent

Exclusion Criteria:

* Coagulation and/or platelets hereditary disorders and/or INR>1.5, PLT<50,000
* Use of anticoagulants that cannot be discontinued
* Pregnant women
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is an observational multicentric prospective study. Data from consecutive patients with AC will be evaluated and, if eligible and agreed to participate, will be recorded in an electronic register. Patients will be followed until death or for at least 1 year after stent removal.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success of EUS-GBD | 2 years
  The rate of successful LAMS placement in the targeted organ
Clinical success of EUS-GBD | 2 years
  The clinical resolution of the Acute cholecystitis

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas-Mater Domini, Castellanza, Italy

IPD SHARING:
Plan to Share IPD: No